CLINICAL TRIAL: NCT06602479
Title: A Phase 2, Randomised, Multicentre, Parallel-Group Treatment, Double-Blind Study to Investigate the Safety and Efficacy of Subcutaneous MEDI0618 in the Reduction of Migraine Headache Days Compared to Placebo in Adult Participants With Episodic Migraine
Brief Title: A Study to Investigate the Safety and Efficacy of MEDI0618 Compared to Placebo in Adult Participants With Episodic Migraine
Acronym: AURORA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D7060C00003; IND 170145 (Registry Identifier: FDA); 2024-512904-21 (Other: EMA)
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: MEDI0618; Episodic Migraine; Migraine headache day(s) - MHD
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: This is parallel-group, participant and investigator blinded, treatment study.
  Approximately 1220 participants will be screened to achieve 488 randomised to study intervention and 438 evaluable participants.
  Study Arms:
  The aCGRP-N cohort includes 5 arms (placebo and 4 active dose levels).
  * A total of 160 participants will be randomised on a 1:1 basis to receive MEDI0618 or placebo.
  * After 104 participants total have been randomised on a 1:1 basis to either MEDI0618 or placebo, 3 other dose arms with MEDI0618 will be initiated and include 56 participants each.
  The aCGRP-IR cohort includes 2 arms (placebo and one active dose level).
  * 2 arms of 80 participants each; 1 will receive MEDI0618 and 1 will receive placebo randomised on a 1:1 basis.
Who Masked: Participant, Investigator
Masking Description: This study will be performed in a double-blind manner (ie, investigator and participant blind). The responsible personnel preparing IP at the site will have access to participants' unblinded treatment assignments.
  The IRT/RTSM will provide to the investigators or pharmacists the kit identification numbers to be allocated to the participant at the dispensing visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- aCGRP-N_MEDI0618 (Dose A) (Experimental): In the aCGRP-N cohort, 160 participants will be randomised on a 1:1 basis to receive MEDI0618 Dose A or placebo.
  After 104 participants total have been randomised, 3 other dose arms with MEDI0618 will be initiated and include 56 participants each.
  Interventions: Drug: MEDI0618
- aCGRP-N_Placebo (Placebo Comparator): In the aCGRP-N cohort, 160 participants will be randomised on a 1:1 basis to receive MEDI0618 Dose A or placebo.
  After 104 participants total have been randomised, 3 other dose arms with MEDI0618 will be initiated and include 56 participants each.
  Interventions: Drug: Placebo
- aCGRP-N_MEDI0618 (Dose B) (Experimental): After 104 participants total have been randomised on Dose A and placebo arms, MEDI0618 will be initiated and include 56 participants each on active dose arm.
  Interventions: Drug: MEDI0618
- aCGRP-N_MEDI0618 (Dose C) (Experimental): After 104 participants total have been randomised on Dose A and placebo arms, MEDI0618 will be initiated and include 56 participants each on active dose arm.
  Interventions: Drug: MEDI0618
- aCGRP-N_MEDI0618 (Dose D) (Experimental): After 104 participants total have been randomised on Dose A and placebo arms, MEDI0618 will be initiated and include 56 participants each on active dose arm.
  Interventions: Drug: MEDI0618
- aCGRP-IR_MEDI0618 (Dose A) (Experimental): In the aCGRP-IR cohort there will be 1:1 randomisation of participants (80 to MEDI0618 and 80 to placebo).
  Interventions: Drug: MEDI0618
- aCGRP-IR_Placebo (Placebo Comparator): In the aCGRP-IR cohort there will be 1:1 randomisation of participants (80 to MEDI0618 and 80 to placebo).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI0618 — MEDI0618 per protocol
  Arms: aCGRP-IR_MEDI0618 (Dose A); aCGRP-N_MEDI0618 (Dose A); aCGRP-N_MEDI0618 (Dose B); aCGRP-N_MEDI0618 (Dose C); aCGRP-N_MEDI0618 (Dose D)
Drug: Placebo — Volume-matched placebo for all arms
  Arms: aCGRP-IR_Placebo; aCGRP-N_Placebo

SUMMARY:
The purpose of this Phase 2 study is to evaluate the safety and efficacy of SC MEDI0618 compared to placebo in participants with episodic migraine.

DETAILED DESCRIPTION:
This Phase 2, randomised, multicentre, parallel-group treatment, double-blind, placebo -controlled study is designed to evaluate the safety and efficacy of subcutaneous (SC) MEDI0618 in participants with episodic migraine.

The study includes a cohort of participants who have a history of unsuccessful treatment with ≥ 2 small molecule migraine preventive treatments from different classes and are eligible to receive an aCGRP therapy (aCGRP-N) but have not yet done so; The study also includes a smaller cohort of participants who have failed one or more aCGRP therapies (aCGRP-IRs) used for preventative treatment and have a history of unsuccessful treatment with ≥ 2 small molecule migraine preventive treatments from different classes.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* Weight ≥ 40 kg and BMI ≥ 18.0 kg/m2.
* History of migraine headaches with or without aura, with migraine onset at ≤ 50 years of age and for at least 12 months prior to screening.
* At least 12 MHDs over the last 3 months prior to screening.
* Participants must fulfil the following criteria for migraine in prospectively collected baseline information during the 4 consecutive weeks of baseline migraine headache data collection prior to Day 1: (a) ≥ 4 and ≤ 14 MHDs per month. (b) On ≥ 4 days, fulfils any of the following criteria: (i) migraine without aura; (ii) migraine with an aura symptom accompanied or followed by a headache within 60 minutes; (iii) probable migraine; (iv) recurrent attacks that do not match ICHD criteria for migraine but successfully respond to migraine-specific medication.
* Participants who fulfil criteria for MOH are eligible for this study.
* History of unsuccessful treatment with ≥ 2 small molecule migraine preventive treatments from different classes (a) aCGRP-N participants are eligible to receive an aCGRP therapy but must have not yet received aCGRP therapy for acute or preventive treatment at any time. (b) aCGRP-IR participants must have tried and have failed at least one aCGRP therapy used for preventive treatment.
* Participants must be able to distinguish migraine headaches from tension-type headaches.
* Female participants who are not pregnant and do not plan to become pregnant during the study, are not lactating, or are of nonchildbearing potential. FOCBP who are sexually active with a non-sterilised male partner must use adequate contraception consisting of two highly effective methods of contraception throughout the study. FOCBP must agree to comply with protocol specified guidance for safe administration of MEDI0618. FOCBP must refrain from egg donation and in vitro fertilisation from the time of signing the ICF, throughout the study, and for 10 weeks after the last administration of investigational product (IP).

Exclusion Criteria:

* History of migraine sub-types including hemiplegic (sporadic or familial) migraine, ophthalmoplegic migraine, and basilar-type migraine
* History of headache other than migraine within 3 months prior to screening.
* History of severe or ongoing allergy/hypersensitivity reactions or history of hypersensitivity to immunisations or immunoglobulins.
* History of any significant psychiatric disorder which could be detrimental to participant safety or could compromise study data interpretation.
* Presence of any clinically significant illness, such as cardiovascular, neurologic (except for non-exclusionary headaches in participants with migraine), pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, or endocrine disease or disorder.
* History of cancer within 5 years of screening, or between screening and randomisation, with the exception of non-metastatic basal cell carcinoma of the skin, carcinoma in situ of the cervix, or non-progressive prostate cancer.
* Known history of drug or alcohol abuse within 1 year of screening or positive test for drugs of abuse or alcohol at screening or at Day -1.
* History of QT prolongation > 450 msec (> 470 msec for participants aged ≥ 65 years) associated with other medications that required discontinuation of that medication.
* Congenital long or short QT syndrome.
* History of arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which is symptomatic or requires treatment, symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication are permitted.
* Use of migraine preventive medications within 30 days or 5 half-lives (whichever is longer) prior to screening and throughout the study
* For aCGRP-N participants only: prior use of an aCGRP therapy for acute or preventive treatment.
* Use of opioids or barbiturate containing analgesic > 2 times/month on average in the 6 months prior to screening for the treatment of pain (opioid administration in an emergency setting may be an exception).
* Use of botulinum toxin (e.g., Botox ®, Dysport®, Jeuveau™, Myobloc®, Xeomin®) for migraine or for any other medical or cosmetic reasons requiring injections in the head, face, or neck during the 4 months prior to screening.
* Use of an intervention or device (eg, scheduled nerve block, transcranial magnetic stimulation) for treatment of migraine within 2 months of screening.
* Use of prescription or non-prescription, non-biologic drugs, including vitamins and herbal and dietary supplements, within 7 days or 5 half-lives (whichever is longer) prior to screening and throughout the study unless the medication will not interfere with the study procedures or compromise participant safety; the dose and regimen must have been stable for at least 3 months prior to screening and must remain stable throughout the study.
* Requires treatment with another biological therapeutic agent including IV immunoglobulin treatment during the course of the study. Prior use of therapeutic antibodies is allowed if that use was > 5 half-lives of the intervention or 3 months prior to screening, whichever is longer.
* Therapeutic vaccines are permitted during the study, but ideally, live attenuated vaccines should be administered > 30 days prior to randomisation and inactivated vaccinations (eg, inactive influenza, COVID-19) should be administered > 14 days prior to randomisation.
* Participation in another clinical study with an IP, including an experimental vaccine, or device, within 5 half-lives of the intervention or 3 months prior to screening, whichever is longer.
* Known hypersensitivity to MEDI0618 or any of the excipients of the product.

Other protocol defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-12-18 (Estimated); Study Completion 2027-05-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of repeat doses of MEDI0618 in preventing migraine headaches in patients with episodic migraine | Week 9 to Week 12
  Change in number of MHDs from 4-week baseline to last 4 weeks of treatment period.

SECONDARY OUTCOMES:
Efficacy of repeat doses of MEDI0618 in preventing migraine headaches in patients with episodic migraine as proportion of patients | Week 9 to Week 12
  Participants with at least 50% reduction in number of MHDs in the last 4 weeks of treatment period compared to 4-week baseline.
Effect of repeat doses of MEDI0618 on disability caused by migraine headaches | Day 1 to Day 85 and to Day 141
  Change in MIDAS score from baseline to end of treatment period and to follow-up.
Effect of repeat doses of MEDI0618 on disability caused by migraine headaches | Day 1, Day 29, Day 57 and Day 85 and to Day 141
  Change in HIT-6 score from baseline throughout the treatment period and to follow-up
Effect of repeat doses of MEDI0618 on the severity of migraine headaches | Week 9 to Week 12
  Change in number of moderate or severe MHDs from 4-week baseline to last 4 weeks of treatment period.
Effect of repeat doses of MEDI0618 on the severity of migraine headaches | Week 9 to Week 12
  Change in number of moderate or severe headache days from 4-week baseline to last 4 weeks of treatment period.
Effect of repeat doses of MEDI0618 on the severity of migraine headaches | Week 9 to Week 12
  Change in frequency of use of permitted acute treatment to abort migraine headaches from 4-week baseline to last 4 weeks of the treatment period.

CONTACTS AND LOCATIONS:
Locations (54):
- United States (16):
  - Flourish - Birmingham, Birmingham, Alabama
  - Tennessee Valley Neurological Associates PC, Huntsville, Alabama
  - The Neurology Center of Southern California - Carlsbad Office, La Jolla, California
  - Clinical Research Institute, LCC, Los Angeles, California
  - Homestead Associates in Research, Inc., Homestead, Florida
  - Florida Neurology - Lake Mary, Lake Mary, Florida
  - Flourish Research - Miami, LLC dba Flourish Research, Miami, Florida
  - BayCare Medical Group Neurology at St. Anthony's Hospital, St. Petersburg, Florida
  - Santos Research Center, Corp - Tampa, Tampa, Florida
  - Norton Neuroscience Institute - Headache Clinic, Louisville, Kentucky
  - Modern Migraine, MD, New York, New York
  - Velocity Clinical Research, Providence (East Greenwich), East Greenwich, Rhode Island
  - Palmetto Primary Care Physicians Division of Gastroenterology - Summerville, Summerville, South Carolina
  - FutureSearch Trials, Austin, Texas
  - Vaught Neurological Services, PLLC, Crab Orchard, West Virginia
  - The Mind+ Neurology Clinic, Mequon, Wisconsin
- Czechia (8):
  - Brain-Soultherapy s.r.o., Kladno
  - Clintrial s.r.o., Prague
  - DADO Medical s.r.o., Prague
  - Axon Clinical s.r.o., Prague
  - Praglandia s.r.o., Prague
  - Forbeli s.r.o, Prague
  - Institut Neuropsychiatricke Pece (INEP), Prague
  - Vestra Clinics s.r.o., Rychnov nad Kněžnou
- Rigshospitalet (Copenhagen University Hospital) - Dansk Hovedpinecenter (Danish Headache Center), Glostrup Municipality, Denmark
- Germany (6):
  - Charite-Universitaetsmedizin Berlin - Campus Charite Mitte (CCM) - Klinik fuer Neurologie, Berlin
  - Pharmakologisches Studienzentrum Chemnitz GmbH, Chemnitz
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Essen, Essen
  - Kopfschmerzzentrum Frankfurt, Frankfurt am Main
  - Fachuebergreifende Gemeinschaftspraxis Dr. med. Joachim Springub & Wolfgang Schwarz, Westerstede
- Hungary (3):
  - Óbudai Egészségügyi Centrum, Budapest
  - S-Medicon Kft., Budapest
  - Obudai Egeszsegugyi Centrum - Dunaujvaros, Dunaújváros
- Italy (4):
  - IRCCS Ospedale San Raffaele, Milan
  - IRCCS Fondazione Istituto Neurologico Nazionale Casimiro Mondino, Pavia
  - Policlinico Universitario Campus Bio-Medico, Roma
  - IRCCS San Raffaele Pisana, Roma
- Poland (10):
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Pratia - Katowice, Katowice
  - Specjalistyczne Gabinety Sp. z o.o., Krakow
  - FutureMeds Sp. z.o.o., Krakow
  - Centrum Medyczne Hope Clinic, Lublin
  - Solumed Centrum Medyczne, Poznan
  - Centrum Medyczne HCP Sp. z o.o., Poznan
  - FutureMeds Warszawa Centrum, Warsaw
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - European Trial Group (ETG) - Warszawa, Warsaw
- Spain (6):
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron - Institut de Recerca (VHIR), Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/